CLINICAL TRIAL: NCT06055894
Title: Microbial Changes in Response to a Plant Based Diet and/or Supplements in SMM/MGUS Patients: A National Multi-Arm Randomized Prospective Telehealth Study Via HealthTree
Brief Title: A Study of a Plant-Based Diet and Dietary Supplements in People With Smoldering Multiple Myeloma (SMM) or Monoclonal Gammopathy of Undetermined Significance (MGUS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: HealthTree Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-116
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma, Smoldering; Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance
Keywords: Plant-Based Diet; Dietary Supplements; 23-116
MeSH Terms: conditions — Smoldering Multiple Myeloma; Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance | interventions — Docosahexaenoic Acids; Curcumin; Probiotics; Diet, Plant-Based

STUDY DESIGN:
Intervention Model Description: This is a randomized, non blinded, telehealth based, national pilot study with 100 patients (25 per arm). Randomization will be stratified based on BMI (normal/elevated) and Mayo risk SMM criteria.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Omega-3 (Experimental): For 2 weeks, patients will receive omega 3 fatty acid supplements 1640 mg (2 capsules) twice daily Qwell™ Omega 3 by The Veggie Doctor™. Each 820 mg omega 3 supplement capsule contains 700 mg Docosohexaenoic acid, 100 mg Docosapentaenoic acid, and 20 mg Eicosapentaenoic acid. No dietary changes will be made but data on dietary intake will be collected.
  Interventions: Dietary Supplement: Omega-3
- Curcumin (Experimental): For 2 weeks, patients in the curcumin arm will receive Curcumin C3 complex 1000 mg with 5 mg BioPerine twice daily from Sabinsa pharmaceuticals. No dietary changes will be made but data on dietary intake will be collected.
  Interventions: Dietary Supplement: Curcumin
- Probiotic (Experimental): For 2 weeks, patients in the probiotic arm will receive Ultra-50 probiotics with 50 billion CFU per capsule (one capsule) twice daily from Vita Miracle pharmaceuticals. No dietary changes will be made but data on dietary intake will be collected.
  Interventions: Dietary Supplement: Probiotic
- Whole food, plant-based diet (WFPBD) (Experimental): For 2 weeks, on the WFPBD arm, patients will receive 14 items weekly, prepared and shipped by U.S. based company, Daily Harvest once a week. The meals will have range from 2 breakfast, 11 lunch/dinners, 1 snack (provided Week 1), and whole grains items (provided Week 2). The meals will contain legumes, fruits, vegetables, whole grains, and plant-based fats that have undergone minimal processing. Detailed recommendations for additional meals outside those given by Daily Harvet meeting the standard of a WFPBD will also be given to supplement their individual daily calorie needs through the guidance of the research dietitian. Patients will receive a varied menu created by Daily Harvest and the study team on a weekly basis.
  Interventions: Other: Whole food, plant-based diet (WFPBD)

INTERVENTIONS:
Dietary Supplement: Omega-3 — For 2 weeks, patients will receive omega 3 fatty acid supplements 1640 mg (2 capsules) twice daily
  Arms: Omega-3
Dietary Supplement: Curcumin — For 2 weeks, patients in the curcumin arm will receive Curcumin C3 complex 1000 mg with 5 mg BioPerine twice daily
  Arms: Curcumin
Dietary Supplement: Probiotic — For 2 weeks, patients in the probiotic arm will receive Ultra-50 probiotics with 50 billion CFU per capsule (one capsule) twice daily
  Arms: Probiotic
Other: Whole food, plant-based diet (WFPBD) — Daily Harvest once a week. The meals will have range from 2 breakfast, 11 lunch/dinners, 1 snack (provided Week 1), and whole grains items (provided Week 2).
  Arms: Whole food, plant-based diet (WFPBD)

SUMMARY:
The researchers are going this to look at how butyrate levels change in participants' stool after they are on a plant-based diet or dietary supplements (omega-3, curcumin or probiotics) for 2 weeks. All participants will have smoldering multiple myeloma (SMM) or monoclonal gammopathy of undetermined significance (MGUS). The researchers will compare how the different dietary changes affect butyrate levels in participants' stool.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed prior diagnosis MGUS or of smoldering myeloma (any time prior). However, confirmation of diagnosis must be documented in their last local oncologist clinic note within 6 months prior to study enrollment.
* Age ≥18 years
* Willingness to comply with all study-related procedures
* Physically able to complete requirements for the study or has someone to assist with the requirements (such as meal preparation, stool shipment and survey completion)
* Interested in learning to cook plant-based recipes
* Access to smart mobile phone or device with camera and ability to download Keenoa app
* Be residing within the United States for the study duration.
* English speaking or a family member or caregiver who speaks English and is able to assist with the surveys and phone based Keenoa app.

Exclusion Criteria:

* Taking any supplements other than vitamin D, iron, vitamin B12, potassium, magnesium, calcium or those needed for a medical indication must be reviewed by PI. If patient is on a supplement (including curcumin, probiotic, omega3) they must stop these for 2 weeks prior to enrollment on study.
* Patients that already follow a whole foods plant based diet (ovo-lactovegetarian or processed junk food vegan diets are not excluded). This will be per research dietitian evaluation and discretion after nutrition screening.
* Legume allergy
* Severe allergies such as anaphylactic shock to peanuts and/or tree nuts, such as cashews
* Concurrent participation in weight loss/dietary trials or defined programs (that require specified diets/supplements on the program). Patients on weight loss drugs are eligible.
* Mental impairment leading to inability to cooperate
* Enrollment onto any other therapeutic investigational study
* Concurrent pregnancy
* Patients on full dose anticoagulation
* If in the opinion of the investigator there maybe any concerns regarding the ability of the patient to complete the study safely
* Current self-reported heavy alcohol use and is defined as >5 drinks per day or >15 drinks per week
* Current self-reported illicit drug use (except inhaled marijuana, vaping or cigarette smoking or medical marijuana.
* Has a condition requiring antibiotics within 14 days of study intervention administration.
* Plan for travel during the study that would preclude adherence to prescribed diets
* History of active inflammatory bowel disease or major gastrointestinal surgery (not including appendectomy or cholecystectomy) within 3 months of enrollment or any history of total colectomy, or bariatric surgery (bariatric surgery which does not disrupt the gastrointestinal lumen, i.e. restrictive procedures such as banding, are permitted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Relative abundance of stool butyrate producers at 2 weeks | at 2 weeks
  To evaluate the change in stool butyrate levels, which is defined as the average of -1 and 0 week samples. Patient stool will be assessed for butyrate levels in batches by gas chromatography mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Urvi A Shah, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm